CLINICAL TRIAL: NCT05670314
Title: Molecular Signatures of Endocannabinoid Induced Pain Relief in Humans: Lifestyle Interventions, Systemic and Localised Changes
Brief Title: lIfestyle iNterventionS for PaIn ReliEf (INSPIRE)
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 22025
Record Dates: First submitted 2022-11-18; First posted 2023-01-04 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — maltodextrin; Exercise

STUDY DESIGN:
Intervention Model Description: 2x2 intervention with individuals per block: placebo (n=27), diet only (n=26), exercise only (n=40), diet + exercise (n=24)
Who Masked: Participant, Investigator
Masking Description: Randomisation will be performed using an online software (sealedenvelope.com). The inulin vs placebo allocation will be double blinded. The exercise part of the intervention will not be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo arm (Placebo Comparator): The participants in the placebo/control arm will be required to take 10g of maltodextrin for the same period of 6 weeks.
  Interventions: Dietary Supplement: Maltodextrin (Placebo)
- Diet only Arm (Experimental): The participants in the dietary intervention arm will be required to take 20g of inulin for a period of 6 weeks.
  Interventions: Dietary Supplement: Inulin Fibre supplement
- Exercise only arm (Experimental): Joint Academy An app-based exercises platform (Joint Academy®) will be used as an intervention given to the treatment arm. The programme consists of a mixture of open and close chain exercises, a combination of concentric, eccentric and focusing on the global strength of legs including the muscles around the hips and knee joints as well as balance enhancement exercises. The intervention also includes educational sessions integrated into the programme covering the basics of OA, its treatment, self-managing symptoms of OA and the benefits of maintaining a healthy lifestyle. The exercise intervention focuses on core stability and performance, neuromuscular leg strengthening and balance enhancement.
  Interventions: Behavioral: Exercise
- Diet + exercise intervention arm (Experimental): The participants in this arm will be required to take 20g of inulin for a period of 6 weeks and doing exercise at the same time.
  Interventions: Dietary Supplement: Inulin Fibre supplement; Behavioral: Exercise

INTERVENTIONS:
Dietary Supplement: Inulin Fibre supplement — 20g/ day. Inulin is easily dissolvable in liquid and can be incorporated into the usual diet - by adding to water, juice, smoothies, cereal, yogurt etc.
  Arms: Diet + exercise intervention arm; Diet only Arm
Dietary Supplement: Maltodextrin (Placebo) — 10g/ day which can be consumed by adding to breakfast cereal/ smoothie/ yogurt or drink of choice
  Arms: Placebo arm
Behavioral: Exercise — Joint Academy An app-based exercises platform (Joint Academy®) will be used as an intervention given to the treatment arm. The programme consists of a mixture of open and close chain exercises, a combination of concentric, eccentric and focusing on the global strength of legs including the muscles around the hips and knee joints as well as balance enhancement exercises.
  Arms: Diet + exercise intervention arm; Exercise only arm

SUMMARY:
This is a 2x2 factorial design randomised controlled trial in which participants with knee pain will be grouped into the diet intervention, exercise intervention, diet and exercise intervention or placebo arm. The study involves intake of dietary supplements and performing routine exercises which are commonly used and are not pharmacological agents. N= 117. 2x2 intervention with individuals per block: placebo (n=27), diet only (n=26), exercise only (n=40), diet + exercise (n=24)

ELIGIBILITY:
Inclusion Criteria:

* Participants with any pain in or around a knee on most days for more than 3 months
* Participant is willing and able to give informed consent for participation in the study
* Participant eligibility includes those aged >18 years who have a body mass index (BMI) between 18.5 and 39.9 kg/m2

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Have psychosocial or gastrointestinal (e.g. malabsorptive conditions such as IBS/IBD, coeliac)
* Are taking the following medications: immunosuppressants, anticoagulants, amiodarone and/or perhexiline
* Are currently following or anticipated to commence a specialised commercially available weight loss diet and/or program
* Pregnant or breast feeding
* History or current psychiatric illness
* History or current neurological condition (e.g. epilepsy)
* Those undergoing revision, having severe hip OA, inflammatory arthropathies
* Diagnosed non-OA cause of knee pain (e.g. rheumatoid arthritis)
* Neuropathy or diabetes mellitus
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance (this must remain for ALL UoN FMHS UREC approved studies)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Valdes, PhD, Principal Investigator — Professor in Genetic and Molecular Epidemiology
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
To comply with the data protection act, personal data will be deleted as soon as possible after it is no longer needed for the study.

REFERENCES:
- [Background] Cui A, Li H, Wang D, Zhong J, Chen Y, Lu H. Global, regional prevalence, incidence and risk factors of knee osteoarthritis in population-based studies. EClinicalMedicine. 2020 Nov 26;29-30:100587. doi: 10.1016/j.eclinm.2020.100587. eCollection 2020 Dec. PMID 34505846
- [Background] Yu D, Peat G, Bedson J, Jordan KP. Annual consultation incidence of osteoarthritis estimated from population-based health care data in England. Rheumatology (Oxford). 2015 Nov;54(11):2051-60. doi: 10.1093/rheumatology/kev231. Epub 2015 Jul 9. PMID 26163287
- [Background] Moseng T, Vliet Vlieland TPM, Battista S, Beckwee D, Boyadzhieva V, Conaghan PG, Costa D, Doherty M, Finney AG, Georgiev T, Gobbo M, Kennedy N, Kjeken I, Kroon FPB, Lohmander LS, Lund H, Mallen CD, Pavelka K, Pitsillidou IA, Rayman MP, Tveter AT, Vriezekolk JE, Wiek D, Zanoli G, Osteras N. EULAR recommendations for the non-pharmacological core management of hip and knee osteoarthritis: 2023 update. Ann Rheum Dis. 2024 May 15;83(6):730-740. doi: 10.1136/ard-2023-225041. PMID 38212040
- [Background] Jonsson T, Eek F, Dell'Isola A, Dahlberg LE, Ekvall Hansson E. The Better Management of Patients with Osteoarthritis Program: Outcomes after evidence-based education and exercise delivered nationwide in Sweden. PLoS One. 2019 Sep 19;14(9):e0222657. doi: 10.1371/journal.pone.0222657. eCollection 2019. PMID 31536554
- [Background] Gohir SA, Eek F, Kelly A, Abhishek A, Valdes AM. Effectiveness of Internet-Based Exercises Aimed at Treating Knee Osteoarthritis: The iBEAT-OA Randomized Clinical Trial. JAMA Netw Open. 2021 Feb 1;4(2):e210012. doi: 10.1001/jamanetworkopen.2021.0012. PMID 33620447
- [Background] Zhang S, Wang D, Zhao J, Zhao H, Xie P, Zheng L, Sheng P, Yuan J, Xia B, Wei F, Zhang Z. Metabolic syndrome increases osteoarthritis risk: findings from the UK Biobank prospective cohort study. BMC Public Health. 2024 Jan 19;24(1):233. doi: 10.1186/s12889-024-17682-z. PMID 38243159
- [Background] Brain K, Burrows TL, Rollo ME, Chai LK, Clarke ED, Hayes C, Hodson FJ, Collins CE. A systematic review and meta-analysis of nutrition interventions for chronic noncancer pain. J Hum Nutr Diet. 2019 Apr;32(2):198-225. doi: 10.1111/jhn.12601. Epub 2018 Oct 7. PMID 30294938
- [Background] Fortuna R, Wang W, Mayengbam S, Tuplin EWN, Sampsell K, Sharkey KA, Hart DA, Reimer RA. Effect of prebiotic fiber on physical function and gut microbiota in adults, mostly women, with knee osteoarthritis and obesity: a randomized controlled trial. Eur J Nutr. 2024 Sep;63(6):2149-2161. doi: 10.1007/s00394-024-03415-w. Epub 2024 May 7. PMID 38713231
- [Background] Woodhams SG, Sagar DR, Burston JJ, Chapman V. The role of the endocannabinoid system in pain. Handb Exp Pharmacol. 2015;227:119-43. doi: 10.1007/978-3-662-46450-2_7. PMID 25846617
- [Background] Ding W, You Z, Chen Q, Yang L, Doheny J, Zhou X, Li N, Wang S, Hu K, Chen L, Xia S, Wu X, Wang C, Zhang C, Chen L, Ritchie C, Huang P, Mao J, Shen S. Gut Microbiota Influences Neuropathic Pain Through Modulating Proinflammatory and Anti-inflammatory T Cells. Anesth Analg. 2021 Apr 1;132(4):1146-1155. doi: 10.1213/ANE.0000000000005155. PMID 32889847
- [Background] Millar B, McWilliams DF, Abhishek A, Akin-Akinyosoye K, Auer DP, Chapman V, Doherty M, Ferguson E, Gladman JRF, Greenhaff P, Stocks J, Valdes AM, Walsh DA. Investigating musculoskeletal health and wellbeing; a cohort study protocol. BMC Musculoskelet Disord. 2020 Mar 21;21(1):182. doi: 10.1186/s12891-020-03195-4. PMID 32199451
- [Background] Karandikar N, Vargas OO. Kinetic chains: a review of the concept and its clinical applications. PM R. 2011 Aug;3(8):739-45. doi: 10.1016/j.pmrj.2011.02.021. PMID 21871418
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Barry E, Galvin R, Keogh C, Horgan F, Fahey T. Is the Timed Up and Go test a useful predictor of risk of falls in community dwelling older adults: a systematic review and meta-analysis. BMC Geriatr. 2014 Feb 1;14:14. doi: 10.1186/1471-2318-14-14. PMID 24484314
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Arant KR, Katz JN, Neogi T. Quantitative sensory testing: identifying pain characteristics in patients with osteoarthritis. Osteoarthritis Cartilage. 2022 Jan;30(1):17-31. doi: 10.1016/j.joca.2021.09.011. Epub 2021 Sep 28. PMID 34597800
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Thorstensson CA, Garellick G, Rystedt H, Dahlberg LE. Better Management of Patients with Osteoarthritis: Development and Nationwide Implementation of an Evidence-Based Supported Osteoarthritis Self-Management Programme. Musculoskeletal Care. 2015 Jun;13(2):67-75. doi: 10.1002/msc.1085. Epub 2014 Oct 24. PMID 25345913
- [Background] Luan L, El-Ansary D, Adams R, Wu S, Han J. Knee osteoarthritis pain and stretching exercises: a systematic review and meta-analysis. Physiotherapy. 2022 Mar;114:16-29. doi: 10.1016/j.physio.2021.10.001. Epub 2021 Oct 11. PMID 35091326

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Started | 27 | 26 | 40 | 24
Completed | 27 | 26 | 40 | 24
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A completers analysis was conducted using the participant numbers shown below.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm | Total
Number analyzed (Participants) | 27 | 26 | 40 | 24 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age (years)
  Years | 69.59 (6.41) | 66.54 (11.39) | 67.75 (10.22) | 66.71 (8.44) | 67.69 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex
  Participants
    Female | 14 | 14 | 26 | 14 | 68
    Male | 13 | 12 | 14 | 10 | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Mean (Standard Deviation); unit: kg/m2] — Body mass index (kg/m2)
  kg/m2 | 29.60 (4.65) | 30.15 (3.75) | 29.00 (7.15) | 29.60 (4.65) | 29.48 (5.32)
Pain Numerical Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Participants reported their pain on a scale ranging from 0 to 10, where 0 represents no pain and 10 indicates the worst pain imaginable
  units on a scale | 3.52 (2.77) | 4.06 (2.85) | 4.21 (2.88) | 3.92 (1.75) | 3.96 (2.67)

OUTCOME MEASURES:

1. Primary Outcome: Change in Numerical Rate Score (NRS) for Pain
Description: The Numerical Rate Score (NRS) will be used to assess the changes in the level of pain in response to the intervention between baseline and follow-up.
  Participants reported their pain on a scale ranging from 0 to 10, where 0 represents no pain and 10 the worst pain imaginable.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 27 | 26 | 40 | 24
units on a scale | 0.67 (2.49) | -0.73 (2.32) | -1.25 (2.69) | -1.21 (1.76)

2. Secondary Outcome: Change in Functional Outcome 30-seconds Sit-to-stand (30CST)
Description: Measures how many times a participant can rise from a chair to a full standing position in 30 seconds.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: stands
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 27 | 26 | 40 | 24
stands | 1.23 (1.67) | 2.12 (3.02) | 2.54 (3.38) | 3.21 (5.37)

3. Secondary Outcome: Change in Functional Outcome Timed-up and go (TUG)
Description: Time in seconds to stand up, walk 3m, return, and sit. Average of 3 trials at baseline and follow-up (at the end of 6 weeks).
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 27 | 26 | 40 | 24
seconds | -0.43 (1.06) | -1.19 (2.19) | -2.07 (5.82) | -0.78 (1.14)

4. Secondary Outcome: Change in Functional Outcome Grip Strength
Description: Measured with dynamometer; average of 3 trials on dominant hand in seated position with participant applying as much grip pressure as possible on the dynamometer. The maximum reading (kg) in taken for each repetition.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 27 | 26 | 40 | 24
kg | -1.43 (6.44) | 0.76 (3.42) | 0.02 (5.62) | 0.76 (3.42)

5. Secondary Outcome: Change in Pain Sensitisation Outcome Temporal Summation (TS)
Description: Pain sensitisation will be measured using quantitative sensory testing (QST) to assess any changes in pain sensitisation indices from at baseline to follow-up. QST is a non-invasive method to assess pain sensitivity using standardised stimuli like mechanical pressure or sharpness. We used the QST modality temporal summation (TS). TS assesses sensitivity to sharpness by applying a brief "pinprick" stimulus (256 mN Pinprick; MRC-Systems, Heidelberg, Germany) to the skin with higher ratings potentially suggesting increased spinal cord pain sensitivity. A single stimulus was applied to the rectus femoris (5cm above the mid-point of the patella of the most painful knee), followed by 10 repetitive stimuli at 1/s. Participants rated pain/sharpness intensity on a 0-10 Visual Analogue Scale after both the single and the average of the repeated stimuli. Each test was performed twice, with a 2-minute break between repetitions and the average was taken.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 27 | 26 | 40 | 24
units on a scale | 0.30 (1.66) | -0.20 (1.52) | -0.17 (1.62) | -0.63 (2.01)

6. Secondary Outcome: Changes in Pain Sensitisation Outcome Pressure Pain Detection Threshold (PPT) at the Superolateral Patella Site
Description: Pain sensitisation will be measured using quantitative sensory testing (QST) to assess any changes in pain sensitisation indices from at baseline to follow-up. QST is a non-invasive method to assess pain sensitivity using standardised stimuli like mechanical pressure or sharpness. We used the QST modality pressure pain detection threshold (PPT) at anatomical position: quadricep (2cm above superolateral edge of patella). PPT measures the lowest pressure a participant perceives as painful while pressure is applied using a handheld probe (Medoc-AlgoMed, Israel) at a rate of 50 kPa/s on the most painful knee, with lower PPT threshold suggestive of increased pain sensitivity.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 27 | 26 | 40 | 24
kPa | -87.19 (103.53) | -29.89 (175.35) | -92.74 (159.03) | -39.22 (240.27)

7. Secondary Outcome: Changes in Pain Sensitisation Outcome Pressure Pain Detection Threshold (PPT) at the Superomedial Patella Site
Description: Pain sensitisation will be measured using quantitative sensory testing (QST) to assess any changes in pain sensitisation indices from at baseline to follow-up. QST is a non-invasive method to assess pain sensitivity using standardised stimuli like mechanical pressure or sharpness. We used the QST modality pressure pain detection threshold (PPT) at anatomical position: quadricep (2cm above superomedial edge of patella). PPT measures the lowest pressure a participant perceives as painful while pressure is applied using a handheld probe (Medoc-AlgoMed, Israel) at a rate of 50 kPa/s on the most painful knee, with lower PPT threshold suggestive of increased pain sensitivity.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 27 | 26 | 40 | 24
kPa | -46.73 (137.77) | -25.33 (122.58) | -41.25 (126.96) | -22.28 (131.10)

8. Secondary Outcome: Changes in Pain Sensitisation Outcome Pressure Pain Detection Threshold (PPT) at the Medial Joint Line Site
Description: Pain sensitisation will be measured using quantitative sensory testing (QST) to assess any changes in pain sensitisation indices from abeline to follow-up. QST is a non-invasive method to assess pain sensitivity using standardised stimuli like mechanical pressure or sharpness. We used the QST modality pressure pain detection threshold (PPT) at the anatomical position: medial joint line (3cm medially from medial edge of patella). PPT measures the lowest pressure a participant perceives as painful while pressure is applied using a handheld probe (Medoc-AlgoMed, Israel) at a rate of 50 kPa/s on the most painful knee, with lower PPT threshold suggestive of increased pain sensitivity.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 27 | 26 | 40 | 24
kPa | -54.54 (132.90) | -31.72 (132.51) | -10.91 (149.56) | -24.02 (160.48)

9. Secondary Outcome: Changes in Pain Sensitisation Outcome Pressure Pain Detection Threshold (PPT) at the Tibialis Anterior Muscle Site
Description: Pain sensitisation will be measured using quantitative sensory testing (QST) to assess any changes in pain sensitisation indices from at baseline to follow-up. QST is a non-invasive method to assess pain sensitivity using standardised stimuli like mechanical pressure or sharpness. We used the QST modality pressure pain detection threshold (PPT) at anatomical position: tibialis anterior (5 cm distal and 1 cm lateral to the tibial tuberosity). PPT measures the lowest pressure a participant perceives as painful while pressure is applied using a handheld probe (Medoc-AlgoMed, Israel) at a rate of 50 kPa/s on the most painful knee, with lower PPT threshold suggestive of increased pain sensitivity.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 27 | 26 | 40 | 24
kPa | -47.36 (160.31) | -17.57 (161.22) | -7.74 (122.59) | -20.66 (180.73)

10. Secondary Outcome: Changes in Pain Sensitisation Outcome Pressure Pain Detection Threshold (PPT) at the Brachioradialis Muscle Site
Description: Pain sensitisation will be measured using quantitative sensory testing (QST) to assess any changes in pain sensitisation indices from baseline to follow-up. QST is a non-invasive method to assess pain sensitivity using standardised stimuli like mechanical pressure or sharpness. We used the QST modality pressure pain detection threshold (PPT) at anatomical position: brachioradialis (5 cm medial and distal to the lateral epicondyle) on the arm opposite the painful knee. PPT measures the lowest pressure a participant perceives as painful while pressure is applied using a handheld probe (Medoc-AlgoMed, Israel) at a rate of 50 kPa/s on the arm opposite the painful knee, with lower PPT threshold suggestive of increased pain sensitivity.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 27 | 26 | 40 | 24
kPa | -27.77 (107.82) | -69.33 (119.04) | -37.31 (95.64) | -25.75 (150.32)

11. Secondary Outcome: Change in Short Chain Fatty Acid Butyric Acid
Description: Change in serum levels of short-chain fatty acid (SCFA) butyric acid in response to the interventions. SCFA levels in serum will be measured using mass spectrometry.
Time Frame: Baseline and 6 weeks
Population: This analysis excludes individuals who either did not provide blood samples or whose values fell below the detection limit and thus did not pass quality control.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 22 | 22 | 25 | 21
ng/ml | -36.67 (1082.93) | 345.61 (434.30) | -233.17 (991.08) | 769.14 (3413.58)

12. Secondary Outcome: Change in Short Chain Fatty Acid Acetic Acid
Description: Change in serum levels of short-chain fatty acid (SCFA) acetic acid in response to theinterventions. SCFA levels in serum will be measured using mass spectrometry.
Time Frame: Baseline and 6 weeks
Population: This analysis excludes individuals who either did not provide blood samples or whose values fell belowthe detection limit and thus did not pass quality control.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 22 | 22 | 25 | 21
ng/ml | -869.59 (3744.05) | 306.32 (1406.99) | -1081.01 (3561.43) | 110.37 (3334.09)

13. Secondary Outcome: Change in Inflammatory Protein Interleukin-6 (IL-6) Levels
Description: Change in Interleukin-6 (IL-6) inflammatory protein levels measured with the Olink for a subset of individuals. For Olink cytokine assay panels data is reported in either Normalized Protein eXpression units (NPX) units or absolute concentration units (pg/mL), with the lower limit of detection typically below 1 pg/mL for most assays.
Time Frame: Baseline and 6 weeks
Population: This analysis excludes individuals who did not provide blood samples or whose values failed quality control or for which results were not obtained
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 3 | 9 | 34 | 23
pg/mL | -1.85 (2.45) | -0.70 (2.12) | -0.25 (0.78) | -0.12 (1.92)

14. Secondary Outcome: Change in Tumor Necrosis Factor (TNF) Inflammatory Protein Levels
Description: Change in Tumor Necrosis Factor (TNF) inflammatory protein levels measured with the Olink for a subset of individuals. For Olink cytokine assay panels data is reported in either Normalized Protein eXpression units (NPX) units or absolute concentration units (pg/mL), with the lower limit of detection typically below 1 pg/mL for most assays.
Time Frame: Baseline and 6 weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 3 | 9 | 34 | 23
pg/mL | -0.52 (1.43) | -0.72 (1.92) | -0.39 (0.80) | -0.34 (1.78)

15. Secondary Outcome: Change in Inflammatory Protein Interferon Gamma (IFN-γ) Levels
Description: Change in Interferon gamma (IFN-γ) inflammatory protein levels measured with the Olink for a subset of individuals. For Olink cytokine assay panels data is reported in either Normalized Protein eXpression units (NPX) units or absolute concentration units (pg/mL), with the lower limit of detection typically below 1 pg/mL for most assays.
Time Frame: Baseline and 6 weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 3 | 9 | 34 | 23
pg/mL | 0.32 (1.72) | 0.04 (2.56) | -0.72 (1.25) | -0.36 (2.56)

16. Secondary Outcome: Changes in Gut Microbiome (Shannon Diversity Index)
Description: The gut microbiome will be measured with shotgun metagenomic sequencing of stool samples and the Shannon Diversity Index will be calculated. The Shannon Diversity Index assesses both the richness (number of different species) and evenness (distribution of individuals among species) within the gut microbiome. A higher Shannon index indicates a more diverse microbiome, while a lower index suggests less diversity.
Time Frame: Baseline and 6 weeks
Population: This analysis excludes individuals who did not provide stool samples or whose values failed quality control or for which results were not obtained
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 2 | 22 | 34 | 22
index | 0.01 (0.26) | -0.07 (0.26) | -0.09 (0.31) | -0.08 (0.33)

17. Secondary Outcome: Change in Serum Endocannabinoid Anandamide (AEA) Levels
Description: Serum levels of Endocannabinoid Anandamide (AEA) will be measured using mass spectrometry in samples collected at baseline and at follow-up (at the end of six weeks). This will help us ascertain the change in levels of Endocannabinoid Anandamide (AEA) in response to the intervention.
Time Frame: Baseline and 6 weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 22 | 23 | 25 | 20
nM | 0.32 (0.82) | 0.05 (0.66) | 0.05 (0.70) | 0.31 (0.77)

18. Secondary Outcome: Change in Serum 2-arachidonoylglycerol (2-AG) Endocannabinoid Levels
Description: Serum levels of 2-arachidonoylglycerol (2-AG) Endocannabinoid will be measured using mass spectrometry in samples collected at baseline and at follow-up (at the end of six weeks). This will help us ascertain the change in levels of 2-arachidonoylglycerol (2-AG) Endocannabinoid in response to the intervention.
Time Frame: Baseline and 6 weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 22 | 23 | 25 | 20
nM | 35.45 (72.07) | 6.28 (44.17) | 37.58 (78.17) | 16.83 (79.10)

19. Secondary Outcome: Changes in Calcium Voltage-gated Channel Subunit alpha1 B Gene Expression Levels Using Transcriptomics on a Subset of Individuals
Description: Transcriptomics will be measured using RNA sequencing of blood samples collected at baseline and at follow-up (at the end of six weeks). RNA was extracted from whole blood, and sequencing libraries were prepared and analysed using standard RNA-seq pipelines.
Time Frame: Baseline and 6 weeks
Population: This analysis was conducted on a subset of samples from the Exercise-only and Diet + Exercise intervention arms, as it was designed to assess the effects of exercise alone, as well as the combined effects of exercise and diet, on gene expression. We specifically examined changes in the expression levels (fold change) of a predefined pain-related gene, calcium voltage-gated channel subunit alpha1 B, between baseline and follow-up.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 10 | 9
fold change | 26.37 (79.60) | 49.50 (140.48)

20. Secondary Outcome: Changes in Solute Carrier Family 12 Member 5 Gene Expression Levels Using Transcriptomics on a Subset of Individuals
Description: as for outcome 19
Time Frame: Baseline and 6 weeks
Population: This analysis was conducted on a subset of samples from the Exercise-only and Diet + Exercise intervention arms, as it was designed to assess the effects of exercise alone, as well as the combined effects of exercise and diet, on gene expression. We specifically examined changes in the expression levels (fold change) of a predefined pain-related gene, solute carrier family 12 member 5, between baseline and follow-up.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 10 | 9
fold change | 14.02 (41.60) | 20.75 (59.51)

21. Secondary Outcome: Changes in Sodium Voltage-gated Channel Alpha Subunit 11 Gene Expression Levels Using Transcriptomics on a Subset of Individuals
Description: Transcriptomics will be measured using RNA sequencing of blood samples collected atbaseline and at follow-up (at the end of six weeks). RNA was extracted from whole blood,and sequencing libraries were prepared and analysed using standard RNA-seq pipelines.
Time Frame: Baseline and 6 weeks
Population: This analysis was conducted on a subset of samples from the Exercise-only and Diet + Exercise intervention arms, as it was designed to assess the effects of exercise alone, as well as the combined effects of exercise and diet, on gene expression. We specifically examined changes in the expression levels (fold change) of a predefined pain-related gene, sodium voltage-gated channel alpha subunit 11, between baseline and follow-up
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Exercise Only Arm | Diet + Exercise Intervention Arm
Number analyzed (Participants) | 10 | 9
fold change | 12.26 (33.70) | 31.97 (90.21)

ADVERSE EVENTS:
Time Frame: Day 1 through Day 42 (daily assessments, 7 days/week)
Arm/Group | Placebo Arm | Diet Only Arm | Exercise Only Arm | Diet + Exercise Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26 | 0/40 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/40 | 0/24
Other Adverse Events (participants affected / at risk) | 0/27 | 10/26 | 0/40 | 13/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=27) | Diet Only Arm (N=26) | Exercise Only Arm (N=40) | Diet + Exercise Intervention Arm (N=24)
Wind and bloating (Gastrointestinal disorders) | 0 (0) | 10 (10) | 0 (0) | 13 (13) — 23 participants reported adverse events related to the inulin intervention (e.g. wind and bloating). No adverse events were reported for all other non-inulin groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT05670314/Prot_SAP_000.pdf